CLINICAL TRIAL: NCT04962581
Title: A Prospective Descriptive Study of the Individualized Capnography of Both Lungs During Single Lung Ventilation With Double-lumen Tube
Brief Title: A Prospective Descriptive Study of the Individualized Capnography of Both Lungs During One-lung Ventilation With Double-lumen Tube
Acronym: EtCO2-DLT
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Jean Bussières, Anesthesiologist, Principal Investigator, Clinical Professor, Laval University
Other Study IDs: 2022-3697, 22100
Record Dates: First submitted 2021-07-05; First posted 2021-07-15 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Thoracic Surgery; Video-Assisted; Double-Lumen Tube; Capnography
Keywords: One lung ventilation; Lung collapse; Capnography; Double lumen tube; DLT; Thoracic surgery; VATS; Video-assisted; Video assisted thoracoscopic surgery
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 : Covidien: This cohort will be monitored with the Covidien capnography, which will be connected to the isolated non-ventilated lung during the whole procedure.
- Group 2: General Électrique: This cohort will be monitored with the General Electrique capnography, which will be connected to the isolated non-ventilated lung during the whole procedure.

SUMMARY:
A prospective descriptive study of the use of an individualized capnography to each lung in the context of one-lung ventilation achieved with a double-lumen tube.

- Pilot project and proof of concept

Brief Summary:

* One study suggests a way to predict possible events of hypoxemia (Sat O2 < 90%) during one lung ventilation (OLV) with the use of two individualized capnography devices on each lung during two-lung ventilation before inducing OLV.
* In addition, a recent presentation in the 2021 Thoracic Anesthesia Symposium suggested possible benefits of the use of a capnography device on the non-ventilated lung in the detection of air leaks around the bronchial cuff.
* The same presentation demonstrated the utility of EtCo2 measurement to determine the achievement of complete lung collapse.

With these previous demonstrations, the use of an individualized capnography for each lung can potentially describe different steps during thoracic surgery. Therefore, a descriptive prospective study on patients that require thoracic surgery with use of a double lumen tube is proposed to verify the feasibility of dual capnography during OLV. The use of two different devices, randomized during our study, will also help to identify the impact of different air aspiration levels on our measures.

Such results will allow to put forward prospective projects to help to optimize OLV during thoracic surgeries.

DETAILED DESCRIPTION:
Thoracic surgery (excluding cardiac surgery) requires lung isolation and one-lung ventilation (OLV) to achieve unilateral lung collapse in order to complete the surgery.

One-lung ventilation requires the use of pulmonary isolation techniques. Two main isolation techniques are used by clinicians: double-lumen tubes (DLT) and bronchial blockers (BB). Bronchial blockers are less used than DLT.

Intra-thoracic interventions and consequently one-lung ventilation, are achieved in a lateral decubitus, with the positioning of the operated hemi-thorax exposed. The most dreaded complication during OLV is hypoxemia, which is defined as the desaturation in the patient's oxygen (SpO2 under 90%). The primary goal of one-lung ventilation is to achieve a rapid and complete lung collapse of the operated lung

Lung collapse is a technique that is well mastered and for which the investigators have contributed significantly regarding its execution in our five of our most recent studies.

Recently, a presentation during the 2021 Thoracic Anesthesia Symposium raised our curiosity regarding the induction of lung collapse (1) This presentation detailed the relevance and possible benefits of adding a capnography on the isolated non-ventilated lung. According to the authors, the capnography of the non-ventilated lung could potentially detect air leaks towards the non-ventilated lung around the bronchial cuff and indicate the occurrence of complete lung collapse.

In addition, an observational study demonstrated the utility of individualized capnography on each lung during thoracic surgery with DLT (2). The measure of the exhaled CO2 gradient between both lungs in a lateral decubitus position before one-lung ventilation could help predict the oxygenation level during the subsequent one-lung ventilation.

The capnography is a tool that is used to monitor continuously the concentration of CO2 that is inhaled and exhaled by intubated patients during general anesthesia (GA). The measures are made with a device that samples a certain quantity of air volume inside a common circuit that ensures the ventilation of both lungs. The sample is taken on a connector that is inserted in the mechanical ventilation circuit. Many companies offer such devices. The intrinsic mechanic is the same although the quantity of volume sampled can vary from one model to another. (50mL/min to 200mL/min)

The use of individualized capnography of each lung seems to present potential benefits during three key moments surrounding one-lung ventilation:

- During the period of time before one-lung ventilation, after the lateral positioning.

* The gradient between the exhaled CO2 of both lungs could predict oxygenation levels during one-lung ventilation.
* During the ventilation of both lungs, the exhaled CO2 is proportional to the blood flow in the pulmonary bed. During the ventilation of both lungs in the lateral decubitus position, the blood flow may vary according to the initial perfusion of both lungs. The effect of gravity caused by the patient's lateral position on the isolated non-ventilated lung's perfusion allows for a better oxygenation. Other factors may also influence the gradient. With that said, oxygenation levels during OLV could be proportional to the difference of exhaled CO2 between both lungs during the lateral decubitus position.

These results could change or conduct during OLV by anticipation of a possible desaturation in oxygen, usually unpredictable.

- During the initiation of the one-lung ventilation

o The capnography is installed on the operated isolated and non-ventilated lung. This could help confirm the quality of the lung isolation and guide our conduct in order to correct inadequate isolation. The quality of the lung isolation depends on the adequate position of the bronchial extremity of the left DLT in the main bronchus. It also depends on the bronchial cuff's seal. In the beginning of OLV, fluctuations in the exhaled CO2 by the isolated non-ventilated lung decrease and flatten. If there is an air leak around the bronchial cuff in the main bronchus, the exhaled CO2 curve will show persistent fluctuations, which would indicate a leak or inadequate seal.

The necessity of correction in the placement of the bronchial cuff and isolation could then be guided by the observation of the exhaled CO2 curve.

- During one-lung ventilation

o During OLV, the capnography installed on the non-ventilation lung could help identify the occurrence of complete lung collapse of the isolated lung. This aspect is an important variable in each of our studies on this subject and is difficultly objectifiable.

The capnography could resolve this problem and help objectively identify total lung collapse.

Hypothesis

Our hypothesis concerning the principal goal of this study is that the measure of the exhaled CO2 of the isolated and non-ventilated lung during thoracic surgery will have specific characteristics for each of the steps described previously.

Our hypothesis concerning our secondary goal is that capnographs that have different levels of aspiration will help us observe distinct exhaled CO2 characteristics.

Goals

Principal: Characterize the measures of exhaled CO2 during different steps of OLV for both lungs (ventilated and non-ventilated).

Secondary: Evaluate the performance and reliability between two devices (high and low level of air aspiration) of capnography on the measure of exhaled CO2 of both lungs during OLV.

Methods

In the context of this study, patients requiring elective thoracic surgeries requiring a OLV will benefit from the addition of an additional capnography on the isolated non-ventilated lung (non-dependent lung) from the anesthetic induction until the achievement of complete collapse of the lung. The investigators will exclude patients in whom a bronchial blocker will be used for OLV.

The information about age, sex, weight, height, VEMS, DLCO and surgical side was collected for all the patients.

The capnography usually used at IUCPQ-UL will be placed on the ventilated lung circuit. The capnography system under study will be installed on the circuit of the non-ventilated lung. The ventilation will be adjusted according to the standards of practice at IUCPQ-UL.

During the study, two capnography machines with different aspiration levels will be evaluated. They will be randomized before the induction of anesthesia, to assess the effectiveness of each of these devices during the different peri-VUP assessment periods. These devices are:

1. - GE Healthcare, CARESCAPE, Respiratory Modules Carbon dioxide (CO2) Sampling rate: 120 ± 20 ml / min
2. - Covidien, CAPNOSTREAM 35. Sampling rate: 50 + - 10 ml / min

The measures of exhaled CO2 for the ventilated and non-ventilated lung will be carried out continuously and will be recorded on the various devices used, then transferred to a laptop computer to be inserted into an Excel file. In addition, the ventilation parameters (respiratory rate, end-tidal volume, 2-lung or single-lung ventilation, FiO2 and PEEP) will also be collected manually. This data will then be retrieved and transferred to the Excel file for further analysis.

Stages of observation

1. Period following induction of anesthetic in the supine position.
2. Period in lateral decubitus

   1. Immediate (ventilation of both lungs)
   2. After the start of the OLV until the opening of the pleura
   3. From the opening of the pleura until achievement of complete collapse of the isolated lung.

When the detection of exhaled CO2 is zero in the non-ventilated lung, which could indicate complete collapse, a photo of the video screen showing an overall view of the lung will be taken in order to qualify the lung collapse at that precise moment.

The description of the lung collapse will be done in this photo, according to our usual criteria by an independent assessor after surgery.

The experimental period should last less than two hours.

Statistics Analysis

This study will require the recruitment of 30 patients divided into 2 groups of 15 subjects. This number was determined based on the analysis of the results of a study published in 2009 by Yamamoto et al (8). The sample size was therefore calculated from the results obtained concerning the exhaled CO2 between the two lungs during lateral decubitus positioning. This is included in our primary assessment goal. It will take a total of 13 patients per group for there to be a statistically significant difference with a p <0.05 and a power of 0.95. Indeed, Yamamoto et al. obtained an exhaled CO2 of 36 ± 5 in the upper lung and 29 ± 5 in the lower lung. The groups for each capnography will be rounded to 15 to obtain a total of 30 patients. If a post-randomization exclusion should occur, the capnography randomization will be transferred to the next subject.

The collected data will first be analyzed in a descriptive manner with graphics in order to interpret fluctuations in exhaled CO2 in the isolated lung. Subsequently, Student's T tests will be carried out in order to compare the values obtained for each measurement time. These comparisons will be made between the different periods and between the different capnographs from the mentioned companies. Finally, the CO2 measures at the time of the picture of the isolated lung will be correlated with the quality of the lung collapse as determined by an independent assessor after the intervention.

Perspective

The investigators hope that the data collected during this research project will allow us to demonstrate the potential benefits of an additional capnograph on the isolated lung during OLV. Promising results from this easy-to-use technology could help predict the onset of hypoxemia in some patients. In addition, the quality of lung isolation could be monitored using this technology. Finally, if the exhaled CO2 is shown to be a potential marker of lung collapse, this will standardize the subjective methodology currently used in the literature in which the lung collapse is indicated by photos or videos of the lung. Such results will allow us to put forward prospective projects already under development within our team.

ELIGIBILITY:
Inclusion Criteria:

* Use of double-lumen tubes for isolation of the lung
* Elective unilateral lung resection (anatomical segmentectomy, lobectomy or pneumonectomy) for lung cancer

Exclusion Criteria:

* Use of bronchial blockers
* IMC above 35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Study population is all patients that require one-lung ventilation thoracic surgery with use of double-lumen tubes.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-07-04 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Characterize the expired CO2 during the different steps in one lung ventilation | During Thoracic Surgery: From intubation to extubation
  Characterize the expired CO2 during the different steps in one lung ventilation for both lungs: the isolated non-ventilated and the ventilated lung

SECONDARY OUTCOMES:
Performance and reliability of two capnography machines on the measure of the expired carbon dioxide | During Thoracic Surgery: From intubation to extubation
  Performance and reliability of two capnography machines ( high and low air aspiration debit) on the measure of the expired carbon dioxide in the isolated and non-ventilated lung during the single lung ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Fortier, Principal Investigator — Laval University
Locations (1):
- Institut de cardiologie et de pneumologie de Québec - Université Laval, Québec, Quebec, Canada

REFERENCES:
- [Background] Kiwakyou L. BJ. Free and Simple Confirmation of Lung Isolation adequacy. [Thoracic Anesthesia Symposium 2021, Poster Presentation #30]. In press 2021
- [Background] Yamamoto Y, Watanabe S, Kano T. Gradient of bronchial end-tidal CO2 during two-lung ventilation in lateral decubitus position is predictive of oxygenation disorder during subsequent one-lung ventilation. J Anesth. 2009;23(2):192-7. doi: 10.1007/s00540-008-0737-9. Epub 2009 May 15. PMID 19444556